CLINICAL TRIAL: NCT03905785
Title: Effectiveness of Parenting Intervention for Improving Child Mental Health: Randomised Single Blind Controlled Trial
Brief Title: Effectiveness of Parenting Intervention for Improving Child Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Balavikasa Educational Academy, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMP/Bala/02189
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Behavior Problem; Conduct Disorders in Children; Mental Health Wellness 1
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting Intervention Group(Samarthan) (Experimental): Parenting intervention was designed as group program, training parents in cognitive-behavioural techniques for managing child's difficult behaviour and issues. Program was focused on parent-child problem solving method and positive interaction.
  Interventions: Behavioral: Samarthan
- Wait list Control group (No Intervention): wait list control group was given no intervention for the trial period. They were offered sam intervention after the intervention was completed in experimental group.

INTERVENTIONS:
Behavioral: Samarthan — Samarthan intervention was designed as group program, training parents in cognitive-behavioural techniques for managing child's difficult behaviour and issues. Program was focused on parent-child problem solving method and positive interaction.
  Arms: Parenting Intervention Group(Samarthan)

SUMMARY:
In this study, effectiveness of a group parenting intervention was assessed in a community setting, for its impact on child behaviour problems and parental mental health.

ELIGIBILITY:
Inclusion Criteria:

* Parents who consented to join the trial
* Children aged 2-8 years
* Mean score on the Eyberg Intensity Scale for clinical issues

Exclusion Criteria:

* Any comorbid psychiatric condition in parents or children
* Substance abuse or diagnosed clinical somatic condition influencing ability to consent or follow intervention

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Child Problem Behaviour | Change from baseline to 8 weeks
  Child problem behaviour was assessed using Eyberg Child Behavior Inventory which evaluates parental report of behavioral problems

SECONDARY OUTCOMES:
General Health Questionnaire | Changes from baseline to 8 weeks
  Parents general health was assessed using General Health questionnaire
Parenting stress | Changes from baseline to 8 weeks
  Parenting Stress Index measured parenting stress
Self-esteem | Changes from baseline to 8 weeks
  Self-esteem in parents were measured using Self-esteem score

CONTACTS AND LOCATIONS:
Overall Officials: Sadhana Sharma, MD, Study Chair — NMP Medical Research Institute, India; Neha Sharma, PhD, Study Director — Warwick Research Services; Nagamani Krishnamurthy, PhD, Principal Investigator — Balavikasa Educational Academy, India
Locations (1):
- Gyansanjeevani, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided